CLINICAL TRIAL: NCT02506361
Title: Evaluation of the Relationship of TOP2α Expression and Effect of Anthracyclines Followed Taxanes or Contains no Taxanes Non Dose-dense Chemotherapy for Breast Cancer: a Prospective, Non-interventional, Multicentre Trail
Brief Title: Evaluation of the Relationship of TOP2α Expression and Effect of Non Dose-dense Chemotherapy for Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: E2014168
Record Dates: First submitted 2015-06-08; First posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer
Keywords: TOP2α; anthracyclines; taxanes; non dose-dense chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a prospective、multicenter、non-comparative interventional case series. 800 breast cancer patients who have already received chemotherapy prior to this study will be enrolled in the group, including 400 patients received the anthracyclines followed taxanes chemotherapy, and the other 400 patients who have received regiments containing no taxanes. Three tumor tissue slices of all the enrolled patients will be collected for TOP2α assay. Meanwhile, 10 years followed-up survey will be conducted. The relationship of TOP2α expression and 5- year or 10-year disease free survival(DFS) and overall survival（OS）will be identified in this study.

DETAILED DESCRIPTION:
800 breast cancer patients who have received chemotherapy prior to this study will be enrolled in the group, including 400 patients received the anthracyclines followed taxanes chemotherapy(Epirubicin 90 mg/m2 d1, Cyclophosphamide 600mg/m2 d1，21days/cycle, 4 cycles, followed by Docetaxel 75mg/m2,d1, 21days/cycle, 4 cycles;or paclitaxel：Epirubicin 90 mg/m2 d1 cyclophosphamide 600mg/m2 d1, 21day/cycle, 4 cycles, followed by paclitaxel 80mg/m2, weekly, 12 wks), and the other 400 patients who have received regiments containing no taxanes (FEC：5-FU 600mg/m2 d1,Epirubicin 90mg/m2 d1, Cyclophosphamide 500mg/m2 d1, 21day/cycle, 6 cycles; or EC: Epirubicin 90mg/m2 d1, Cyclophosphamide 500mg/m2 d1,21 day/cycle, 6 cycles).The patients will be enrolled in the groups within one month after chemotherapy.Three tumor tissue slices of all the enrolled patients will be collected for TOP2α assay. Meanwhile, 10 years followed-up survey will be conducted. The relationship of TOP2α expression and 5-year or 10-year disease free survival(DFS) and overall survival（OS）will be identified in this study.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, subjects must fulfil all of the following criteria:

1. . Signed and dated informed consent indicating that the patient (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to enrollment.
2. . Invasive breast cancer confirmed by histology or cytology with the tumor complete resection.
3. . Patients without remote organs metastasis.
4. . The Ages of patients ≥ 18 years and ≤70 years.
5. . Patients with positive axillary lymph nodes, or negative axillary lymph nodes plus one of these conditions: Triple-negative breast cancer, HER- 2(+),Ki-67≥15%.
6. . The values of aspartate aminotransferase(AST),alanine aminotransferase(ALT), alkaline phosphatase(ALP), total bilirubin(TBIL), UREA, CREA were less than 2 times of upper limits of normal at the beginning of aromatase inhibitors（AIs） therapy.
7. . TOP2α is available to be detected in the primary tumour tissue.
8. . Patients received the regimens of anthracyclines followed Taxanes or containing no Taxanes non-dose dense chemotherapy suggested by the guidelines of National Comprehensive Cancer Network （NCCN) 2014.

Exclusion Criteria:

Any of the following is regarded as a criterion for exclusion from the study:

1. . Patients is in the period of pregnancy or lactation.
2. . Bilateral breast cancer, inflammatory breast cancer or carcinoma in situ.
3. . Previous received neo-adjuvant therapy, including chemotherapy, radiotherapy or endocrinotherapy.
4. . Presence of other life-threatening cancers.
5. . Any severe concomitant condition: uncontrolled cardiac disease or uncontrolled diabetes mellitus. et al.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 800 breast cancer patients who have already received chemotherapy prior to this study will be enrolled in the group, including 400 patients who have received the anthracyclines followed taxanes chemotherapy, and the other 400 patients have received regiments containing no taxanes.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2015-05; Primary Completion 2025-05 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
TOP2αexpressions of participants | one year
  The TOP2αexpression levels of the 800 enrolled patients tissue samples will be assayed by immunohistochemistry

SECONDARY OUTCOMES:
Disease Free Survival time of participants | ten year
  Ten years followed-up survey will be conducted to identify the 5-year and 10-year Disease Free Survival time of participants.
Overall Survival time of participants | ten year
  Ten years followed-up survey will be conducted to identify the 5-year and 10-year Overall Survival time of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Zhang, Pro., Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Jin Zhang, Tianjin, China